CLINICAL TRIAL: NCT00607529
Title: Clinical Evaluation of an Investigational Blood Creatinine Point-of-Care Test Device
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Nova Biomedical Corporation (Industry)
Responsible Party: Martin Fleisher, PhD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 07-023
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Cancer
Keywords: Multiple Diseases
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood

GROUPS / COHORTS (1):
- 1: Patients having a creatinine drawn
  Interventions: Other: hand-held POC creatinine analyzer-blood test

INTERVENTIONS:
Other: hand-held POC creatinine analyzer-blood test — This study will require the collection of a finger-puncture capillary blood specimen in addition to one green stoppered heparin containing collection tube. This is taken pre-therapy. The capillary whole blood specimen will be used to perform a creatinine determination on the "investigational" hand-held creatinine analyzer using special test strips for the analysis.

SUMMARY:
This study is being done to see if the Nova Creatinine Meter can give a correct measure of creatinine (a blood test used to measure kidney function) when the blood is taken from a capillary (smallest type of blood vessels). The Nova Creatinine Meter is a hand held device that can be used in a clinic to measure creatinine in about 50 seconds. Current laboratory creatinine testing can take up to an hour. Since chemotherapy patients need to have their creatinine measured prior to treatment, this meter could make testing easier and faster.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Must have a creatinine > or = to than 3.5 mg/dl

Exclusion Criteria:

* Patients who are less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC patients
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary outcomes would be, reduced wait time and increased patient satisfaction. | conclusion of the study

SECONDARY OUTCOMES:
reduced blood loss | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fleisher, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org